CLINICAL TRIAL: NCT01966562
Title: Psychological Well Being, Proactive Attitude and Happiness Effects of Whole-body Vibration vs. Multi-component Training in Aged Women: a Randomized Controlled-trial Study Protocol
Brief Title: PAHA Study: Psychological Active and Healthy Ageing
Acronym: PAHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergamo (Other)
Responsible Party: Principal Investigator, Angelo Compare, Professor, University of Bergamo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCT002899231
Record Dates: First submitted 2013-10-08; First posted 2013-10-21 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-09

CONDITIONS: Aged

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- WBV TRAINING (Experimental): WHOLE-BODY VIBRATION TRAINING
  Interventions: Behavioral: WHOLE-BODY VIBRATION TRAINING
- MC TRAINING (Active Comparator): MULTICOMPONENT TRAINING
  Interventions: Behavioral: MULTICOMPONENT TRAINING
- CG (No Intervention): Control group

INTERVENTIONS:
Behavioral: WHOLE-BODY VIBRATION TRAINING — The vibration stimulus consisted of uniform vertical oscillations Power Plate® Next Generation (Power Plate North America, Northbrook, IL, USA). Subjects stood on the platform holding an quarter squat positions with the feet shoulder-width apart. Then, they perform ankle extensions with the following work sequence (establishing a rhythm of 100 b.p.m.: 1 b.p.m for the concentric phase; and 5 b.p.m. for the eccentric phase). After the familiarization 2-weeks, subjects trained 3 days per week for 6-months (72 sessions) using a vibrating training program that began with 5 sets and a frequency of 35 Hz per session and increasing by 11 sets and 40 Hz frequency the last month maintaining a series of parameters: vibration amplitude (4 mm) working time (60 s) and recovery time (60 s).
  Arms: WBV TRAINING
Behavioral: MULTICOMPONENT TRAINING — This training combined vertical jumps and high intensity walking. During the first month, small reactive vertical jumps (without knee and ankle flexion) were performed. After the first month, subjects performed drop jumps progressively starting at a height of 5 cm and finishing at 25 cm at the end of the programme (increases of 5 cm each month). Additionally, the sets were increased from 4x10 jumps to 6x10 each week, finishing the last week with 4x10. In this sense, the drop jumps were the same each month but the total load (imposed by height) increased progressively. Regarding the aerobic exercise, the load increased progressively along the 6 months. The intensity ranged between 50-75% of reserve heart rate, the volume ranged between 30-60 min.
  Arms: MC TRAINING

SUMMARY:
The PAHA study is a three-arm randomized controlled clinical trial (RCT). The aim of this RCT is to compare the effectiveness of the WHOLE-BODY VIBRATION (WBV) with the Multi-component training control group and control group (CG) for psychological well being, quality of life, proactive attitude and happiness in female aged subjects.

DETAILED DESCRIPTION:
A recent review has moreover suggested that the content (the mental and physical demand or challenge, and the behavioral aspects of the activity) and the context (the social context) of activities are key elements when distinguishing various types. Social activity affects wellbeing or survival by reducing the risks of social isolation and by supplying emotional intimacy, socio-emotional support, reinforcement for one's self-concept and social roles, and the sense of being valued. On the other hand, productive activity may influence health and wellbeing through satisfaction with outcomes, economic gains, mental stimulation, comforting personal routines, sense of purpose, and increased self-efficacy or self-esteem. There are significant relationships between QoL and attitudes toward aging in older adults. It has been in fact demonstrated that a proactive attitude (i.e., exercise, planning ahead, and marshaling support) influences QoL outcomes (i.e., depressive symptomatology and social activities).

Evidence has moreover shown that exist gender differences in engage physical activities and in mood state in ageing. In fact, aged women are less engaged in physical activity than men, probably due to menopausal transition (MT) state. Literature has suggested that women who experience longer MT and increased symptoms have higher stress and increased risk of depression , that in turn may affect their engagement in physical activities.

Starting from current literature, we hypothesize that specific physical activity, WBV, may promote psychological well being and quality of life in female aged subjects. Moreover and therefore, we assume an improvement in proactive attitude and happiness when compared to and Multi-component training control group.

ELIGIBILITY:
Inclusion Criteria:

* Women;
* Age ranged between 55-75 years old.

Exclusion Criteria:

* Male sex;
* Age lower than 55 years old;
* Present levels of DMO lower than 70 g/cm2;
* Being treated for a disease that can affect bone structure or neuromuscular system;
* Have orthopedic prosthetic implants in the lower limbs and / or spine; Have herniated discs;
* Suffer ocular diseases that affect the retina;
* Suffer severe cardiovascular diseases;
* Have a pacemaker, or osteosynthesis material;
* Severe mental illness (active psychosis/suicide risk/severe dementia);
* Linguistic limitations (such as stuttering/untreated audio impairment);
* A significant functional problem (such as unconsciousness/connection to respiration device/confinement to a wheelchair or bed/severe walking disability/need of help with basic daily activities), major depression, anxiety according to DSM-IV criteria.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Psychological General Well-Being Index (PGWBI) | Within one year after the treatment
  The PGWBI. It is a self-administered test with 22 items that assess the subjective sensation of psychological wellbeing. It has been divided in 6 categories: anxiety, depression, self-control, positivity and wellbeing, health and vitality (Grossi et al., 2006).

SECONDARY OUTCOMES:
Subjective Happiness Scale (SHS) | Within one year after the treatment
  It 4-item scale for assessing subjective happiness. Two items ask respondents to characterize themselves using both absolute ratings and ratings relative to peers, whereas the other two items offer brief descriptions of happy and unhappy individuals and ask respondents the extent to which each characterization describes them. The SHS has been validated in 14 studies with a total of 2,732 participants. Preliminary results have indicated that the SHS has high internal consistency, which has been found to be stable across samples. Test-retest and self-peer correlations have suggested good to excellent reliability, and construct validation studies of convergent and discriminant validity have confirmed the use of this scale to measure the construct of subjective happiness (Lyubomirsky & Lepper, 1999).
Proactive Attitude Scale (PA) | Within one year after the treatment
  It assess the presence of a Proactive Attitude that is a relatively persistent personal belief in the rich potential of changes that can be made to improve oneself and one's environment. The proactive attitude has implications for motivation and action. This includes various facets such as resourcefulness, responsibility, values and vision. The psychological construct of Proactive Attitude (PA) present a correlation of r = .56 with general self-efficacy (Schwarzer, 1999)
SF-12 Health Survey | Within one year after the treatment
  It is a self-administered test that assesses the global health status by the subjective point of view of the subject. It has been divided into two principal subscales: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). In particular, it allows to asses concept concerning health, physical functions, pain, general health, vitality, social functioning, emotional functioning and mental health (Kodraliu et al., 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Compare, Ph.D., Principal Investigator — University of Bergamo
Locations (1):
- University of Bergamo, Bergamo, Italy

REFERENCES:
- [Derived] Marin-Cascales E, Rubio-Arias JA, Alcaraz PE. Effects of Two Different Neuromuscular Training Protocols on Regional Bone Mass in Postmenopausal Women: A Randomized Controlled Trial. Front Physiol. 2019 Jul 10;10:846. doi: 10.3389/fphys.2019.00846. eCollection 2019. PMID 31354513
- [Derived] Compare A, Zarbo C, Marin E, Meloni A, Rubio-Arias JA, Berengui R, Grossi E, Shonin E, Martini G, Alcaraz PE. PAHA study: psychological active and healthy aging: psychological wellbeing, proactive attitude and happiness effects of whole-body vibration versus Multicomponent Training in aged women: study protocol for a randomized controlled trial. Trials. 2014 May 20;15:177. doi: 10.1186/1745-6215-15-177. PMID 24886107